CLINICAL TRIAL: NCT01414062
Title: Cocinar Para su Salud! (Cook for Your Life!): Implementing Dietary Change Among Hispanic Breast Cancer Survivors
Brief Title: Cook for Your Life!: Implementing Dietary Change Among Hispanic Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Dawn L. Hershman, Professor, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAE9701; 1R21CA152903-01 (NIH)
Record Dates: First submitted 2011-08-03; First posted 2011-08-11 (Estimated); Results first posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Healthy meals; Cocinar; Dietary; Dietary Intervention; fruits and vegetables; Cancer survivor; Nutrition
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Active Comparator): Participants receiving written dietary recommendations for breast cancer survivors (control arm)
  Interventions: Behavioral: Written dietary recommendations
- Arm B (Experimental): Participants attending Cocinar Para Su Salud Program held over a 12-week period
  Interventions: Behavioral: Cocinar Para Su Salud Program

INTERVENTIONS:
Behavioral: Cocinar Para Su Salud Program — A series of 9 Cocinar Para Su Salud intervention sessions held over a 12-week period. The 12-week intervention period will be divided into 3 groups: motivation, action, and environment. Each topic will use a nutrition roundtable, food shopping field trip, and a cooking class to teach pertinent points, in order to enable participants to progress from the precontemplation, contemplation, and preparation stages of change to the action and maintenance stages.
  Other Names: ¡Cocinar para su salud!
  Arms: Arm B
Behavioral: Written dietary recommendations — Standard of care: one on one meetings with study staff to receive compiled written information on dietary recommendations for breast cancer survivors produced by the New York City (NYC)-based not-for-profit, God's Love We Deliver
  Arms: Arm A

SUMMARY:
The primary objectives of this study are to determine the effect of the dietary intervention (Cocinar para su salud! Program) vs. control (standard written nutrition education materials for cancer survivors) in Hispanic breast cancer survivors with early stage breast cancer on 1) daily servings of fruit and vegetable intake from baseline to 6 months; and 2) percent energy from fat and fat-related dietary habits from baseline to 6 months.

DETAILED DESCRIPTION:
Hispanic women are 20% more likely to die of breast cancer than non Hispanic white women who are diagnosed at a similar age and stage. One reason for this disparity may be differences in post diagnosis dietary behaviors. In order to reduce this disparity, and to improve overall survivorship, culturally appropriate dietary interventions that teach women how to eat a diet high in fruits and vegetables and low in saturated fat need to be developed for Hispanic breast cancer survivors. The investigators propose to conduct a randomized controlled study (n=70, 35 per arm) to test the effects of the ¡Cocinar para su salud! program on changing dietary behaviors among Hispanic breast cancer survivors who have recently completed treatment. The ¡Cocinar para su salud! program is a 12 week course that provides hands on education and instruction in nutrition education, meal preparation, and food shopping in a group setting. All participants will be followed for a total of 12 months, have clinical assessments at baseline, 6 months, and 12 months, and monthly telephone contacts using motivational interview techniques.

ELIGIBILITY:
Inclusion Criteria:

* Female.
* Age 21 years or greater. Both pre- and postmenopausal women will be included in this study. Postmenopausal status will be defined as the absence of menses for > 12 months, serum follicle stimulating hormone (FSH)> 20 milli-international units per milliliter (mIU/ml), or history of bilateral oophorectomy.
* Hispanic descent and fluent in Spanish.
* History of histologically-confirmed stage 0, I, II, or III invasive breast carcinoma without evidence of disease recurrent or metastatic disease at trial entry.
* Minimum of 3 months since last chemotherapy, biologic therapy (i.e., trastuzumab), radiation therapy, and/or breast surgery. Current use of hormonal therapy is permitted.
* No uncontrolled diabetes mellitus, defined as Hgb A1C >7.
* No uncontrolled comorbidities (i.e., hypertension).
* Currently a non-smoker (rationale: women who smoke are much less likely to engage in healthy lifestyle behaviors, and it is probably more important for these women to stop smoking than it is to change their dietary patterns).
* Consumes <5 servings of fruits and vegetables per day, as assessed by the Block Fruit and Vegetable Screener.
* In the pre-contemplation, contemplation, or preparation stage of increasing daily fruit and vegetable intake.
* Access to functional home phone or cell phone.
* Willing and able to participate in all study related activities, including study clinic visits, phone interviews, and nutrition counseling sessions.
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Evidence of recurrent or metastatic breast cancer.
* Uncontrolled diabetes (type 1 or 2), defined as Hemoglobin (Hgb) A1C >7.
* Uncontrolled or significant co-morbid illness including, but not limited to, active or serious infection requiring intravenous antibiotics; symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia; active gastrointestinal bleeding; active liver disease; active malignancy, except for squamous cell carcinoma of the skin, basal cell carcinoma of the skin, carcinoma in situ, Stages Ia or Ib invasive squamous cell carcinoma of the cervix treated by surgery and/or radiation therapy, Stage Ia Grade 1 adenocarcinoma of the endometrium treated with surgery; patients receiving active chemotherapy or radiotherapy; or psychiatric illness/social situations that would limit compliance with study requirements.
* Previously participated in Cook For Your Life! classes.
* Currently active in a dietary change program.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Hershman, MD, MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hooper L, Abdelhamid AS, Jimoh OF, Bunn D, Skeaff CM. Effects of total fat intake on body fatness in adults. Cochrane Database Syst Rev. 2020 Jun 1;6(6):CD013636. doi: 10.1002/14651858.CD013636. PMID 32476140
- [Derived] Shi Z, Richardson JM, Aycinena AC, Gray HL, Paul R, Koch P, Contento I, Gaffney AO, Greenlee H. Psychosocial mediators of dietary change among Hispanic/Latina breast cancer survivors in a culturally tailored dietary intervention. Psychooncology. 2018 Sep;27(9):2220-2228. doi: 10.1002/pon.4799. Epub 2018 Jul 25. PMID 29904989

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 82 participants were enrolled and 12 withdrew, resulting in 70 participants being randomized.
Groups:
- Arm A (Control): Participants receiving written dietary recommendations for breast cancer survivors (control arm)
  Written dietary recommendations: Standard of care: one on one meetings with study staff to receive compiled written information on dietary recommendations for breast cancer survivors produced by the New York City-based not-for-profit, God's Love We Deliver
- Arm B (Cocinar Para Su Salud Program): Participants attending Cocinar Para Su Salud Program held over a 12-week period
  Cocinar Para Su Salud Program: A series of 9 Cocinar Para Su Salud intervention sessions held over a 12-week period. The 12-week intervention period will be divided into 3 groups: motivation, action, and environment. Each topic will use a nutrition roundtable, food shopping field trip, and a cooking class to teach pertinent points, in order to enable participants to progress from the precontemplation, contemplation, and preparation stages of change to the action and maintenance stages.
Period: Overall Study
Arm/Group | Arm A (Control) | Arm B (Cocinar Para Su Salud Program)
Started | 36 | 34
Completed | 31 | 30
Not Completed | 5 | 4
Not completed — Lost to Follow-up | 3 | 2
Not completed — Left Country | 1 | 1
Not completed — Family Disapproval | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm A: Participants receive written dietary recommendations for breast cancer survivors (control arm)
  Written dietary recommendations; Standard of care: one on one meetings with study staff to receive compiled written information on dietary recommendations for breast cancer survivors produced by the NYC-based not-for-profit, God's Love We Deliver
- Arm B: Participants attend the Cocinar Para Su Salud Program held over a 12-week period
  Cocinar Para Su Salud Program: A series of 9 Cocinar Para Su Salud intervention sessions held over a 12-week period. The 12-week intervention period will be divided into 3 groups: motivation, action, and environment. Each topic will use a nutrition roundtable, food shopping field trip, and a cooking class to teach pertinent points, in order to enable participants to progress from the precontemplation, contemplation, and preparation stages of change to the action and maintenance stages.
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 36 | 34 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (10.1) | 55.1 (9.1) | 56.6 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 34 | 70
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 11 | 7 | 18
  White | 14 | 14 | 28
  Native American | 0 | 2 | 2
  Mixed | 6 | 5 | 11
  Colombian | 1 | 0 | 1
  Cuban | 1 | 0 | 1
  Dominican | 30 | 24 | 54
  Ecuadorian | 1 | 4 | 5
  El Salvadorian | 0 | 1 | 1
  Honduran | 1 | 0 | 1
  Mexican | 0 | 1 | 1
  Puerto Rican | 2 | 3 | 5
  Missing Race | 5 | 6 | 11
  Other Ethnicity (not specified) | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36 | 34 | 70

OUTCOME MEASURES:

1. Primary Outcome: Change in Daily Servings of Fruits and Vegetables
Description: The change in participants intake and fruits and vegetables at 6 months (compared to baseline) as determined by diet recalls collected by an interviewer administered questionnaire.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: daily servings of fruits and vegetables
Groups:
- Arm A (Control Arm): Participants receiving written dietary recommendations for breast cancer survivors (control arm)
  Written dietary recommendations: Standard of care: one on one meetings with study staff to receive compiled written information on dietary recommendations for breast cancer survivors produced by the NYC-based not-for-profit, God's Love We Deliver
Arm/Group | Arm A (Control Arm) | Arm B (Cocinar Para Su Salud Program)
Number analyzed (Participants) | 31 | 30
daily servings of fruits and vegetables | -0.1 (0.5) | 2.0 (0.5)

2. Secondary Outcome: Change in Daily Servings of Fruits and Vegetables
Description: The change in participants intake and fruits and vegetables at 12 months (compared to baseline) as determined by diet recalls collected by an interviewer administered questionnaire.
Time Frame: Baseline and 12 months
Population: Data on daily servings of fruits and vegetables were collected from 29 participants from each arm.
Measure: Mean (Standard Deviation); unit: daily servings of fruits and vegetables
Arm/Group | Arm A (Control Arm) | Arm B (Cocinar Para Su Salud Program)
Number analyzed (Participants) | 29 | 29
daily servings of fruits and vegetables | -0.2 (2.5) | 1.6 (2.2)

3. Secondary Outcome: Change in Molecular Biomarkers Associated With Breast Cancer Risk
Description: Fasting blood will be collected at baseline and 12 months to determine whether the change in diet changes participants' biomarkers. Specifically, the change in DNA methylation (a chemical reaction in the body in which a small molecule called a methyl group gets added to DNA) will be measured against the increase in dietary factors.
Time Frame: Baseline and 12 months
Population: Blood samples for DNA methylation were collected for 24 and 23 participants in Arm A and B respectively resulting in 24 (Arm A) and 23 (Arm B) analyzed.
Measure: Mean (Standard Deviation); unit: percentage change in DNA methylation
Groups:
- Arm A (Control): Participants receiving written dietary recommendations for breast cancer survivors (control arm)
  Written dietary recommendations: Standard of care: one on one meetings with study staff to receive compiled written information on dietary recommendations for breast cancer survivors produced by the NYC-based not-for-profit, God's Love We Deliver
Arm/Group | Arm A (Control) | Arm B (Cocinar Para Su Salud Program)
Number analyzed (Participants) | 24 | 23
percentage change in DNA methylation | -0.7 (3.8) | 1.2 (3.5)

4. Secondary Outcome: Change in Weight
Description: The change in weight from baseline to 12 months.
Time Frame: Baseline and 12 months
Population: Data on weight were collected from 29 participants from each arm.
Measure: Mean (Standard Error); unit: kg
Arm/Group | Arm A (Control Arm) | Arm B (Cocinar Para Su Salud Program)
Number analyzed (Participants) | 29 | 29
kg | 2.3 (2.6) | -2.2 (2.6)

5. Secondary Outcome: Change in Body Mass Index (BMI)
Description: The change in BMI from baseline to 12 months.
Time Frame: Baseline and 12 months
Population: Data on BMI were collected from 29 participants from each arm.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Arm A (Control Arm) | Arm B (Cocinar Para Su Salud Program)
Number analyzed (Participants) | 29 | 29
kg/m^2 | -0.6 (2.4) | -1.0 (3.2)

ADVERSE EVENTS:
Time Frame: Data was collected at the following time periods: 3 months, 6 months, and 1 year.
Arm/Group | Arm A (Control) | Arm B (Cocinar Para Su Salud Program)
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30
Other Adverse Events (participants affected / at risk) | 0/31 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes